CLINICAL TRIAL: NCT06283680
Title: The Effect of Nutritional Status and Body Mass Index on Lung Capacity, Functional Capacity and Mortality in End-Stage Lung Patients on the Lung Transplant List
Brief Title: The Effect of Nutrition and BMI on on Lung Capacity, Functional Capacity and Mortality in End-Stage Lung Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Aylin Seylam Küşümler (Other)
Collaborators: Koşuyolu Yüksek İhtisas Training and Research Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Aylin Seylam Küşümler, Assistant Professor, Okan University
Organization: Okan University (Other)
Other Study IDs: 2024
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Lung Transplant
MeSH Terms: interventions — Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Ex patients on the lung transplant waiting list
  Interventions: Procedure: Lung transplantation
- Group 2: Tansplant patients
  Interventions: Procedure: Lung transplantation
- Group 3: Patients waiting on the current list
  Interventions: Procedure: Lung transplantation

INTERVENTIONS:
Procedure: Lung transplantation — Three different groups will be investigated with respect to the effect of NRI, BMI and body fat, muscle ratio on functional capacity, lung capacity, exercise capacity index, all-cause mortality, post-transplant intensive care unit stay and survival time in end-stage lung patients on the lung transplant list.

SUMMARY:
The aim of this study was to investigate the effect of nutritional risk index, BMI and body fat, muscle ratio on functional capacity, lung capacity, exercise capacity index, all-cause mortality, post-transplant intensive care unit stay and survival time in end-stage lung patients on the lung transplant list.

DETAILED DESCRIPTION:
This study aimed to determine the nutritional status of patients awaiting lung transplantation and examine the effects of nutritional status, immunonutrition use, and BMI on lung capacity, mortality, and health status after lung transplantation. The study was designed in two different periods. The first period was a retrospective descriptive study. During this study, we will examine the retrospective nutritional status of patients who are waiting for lung transplantation, those who exited while on the list, or those who have received lung transplantation. In the second phase, we will conduct face-to-face interviews with patients on the lung transplant list, take bioelectrical impedance analyses (BIA), and record 24-hour food consumption to examine their detailed nutritional status.

ELIGIBILITY:
Inclusion Criteria:

1. End-stage lung disease
2. To be on the Lung Transplant list.
3. Being between the ages of 19-65
4. Not having severe psychiatric illness
5. Being fed orally
6. Volunteering to participate in the study for Patients Waiting on the Transplant List

Exclusion Criteria:

1. To be removed from the Lung Transplant List
2. Being pregnant or lactating
3. Severe psychiatric illness
4. Peg or Jeg feeding (unable to feed orally)
5. Missing data in the file

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study consisted of patients who applied to the lung transplantation outpatient clinic at Koşuyolu High Specialised Training and Research Hospital between 2016 and 2022, were listed, were waiting on the list, died while on the list, and received lung transplantation, and met the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
BMI | For one month period
  BMI values are evaluated for the patients for patients waiting on the transplant list, transplanted and exited.

SECONDARY OUTCOMES:
Nutrition risk index | For one month period.
  BMI values are evaluated for the patients for patients waiting on the transplant list, transplanted and exited.

CONTACTS AND LOCATIONS:
Locations (1):
- OkanU, Istanbul, Turkey (Türkiye)